CLINICAL TRIAL: NCT01249820
Title: Pharmacokinetics of Anidulafungin Given Intravenously as Antifungal Prophylaxis to Recipients of an Allogeneic Haematopoietic Stem Cell Transplant Following Myeloablative Chemotherapy or Patients Receiving Intensive Chemotherapy for AML-MDS
Brief Title: Pharmacokinetics of Anidulafungin (Ecalta ®) Intravenous Given to Patients at High Risk for Developing Invasive Fungal Disease
Acronym: ANIDULAPK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UMCN-AKF 10.01 / SC25
Record Dates: First submitted 2010-08-23; First posted 2010-11-30 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Leukemia; Myelodysplastic Syndrome; Leukemia, Myeloid, Acute
Keywords: anidulafungin; antifungal prophylaxis; allogeneic haematopoietic stem cell transplant; myeloablative chemotherapy; AML-MDS; pharmacokinetics
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Anidulafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group A (Experimental): Day 1-15: anidulafungin 200 mg q48h IV maintenance dose (8 dosages)
  Interventions: Drug: anidulafungin 200 mg q48h
- group B (Experimental): Day 1-13: anidulafungin 300 mg q72h IV maintenance dose (5 dosages)
  Interventions: Drug: anidulafungin 300 mg q72h

INTERVENTIONS:
Drug: anidulafungin 200 mg q48h — Day 1-15: anidulafungin 200 mg q48h IV maintenance dose (8 dosages)
  Other Names: Ecalta
  Arms: group A
Drug: anidulafungin 300 mg q72h — Day 1-13: anidulafungin 300 mg q72h IV maintenance dose (5 dosages)
  Other Names: Ecalta
  Arms: group B

SUMMARY:
The purpose of this study is to study the pharmacokinetics of anidulafungin (Ecalta ®) given intravenously as antifungal prophylaxis to recipients of an allogeneic haematopoietic stem cell transplant following myeloablative chemotherapy or patients receiving intensive chemotherapy for AML-MDS who are at high risk for developing invasive fungal disease.

DETAILED DESCRIPTION:
Alternate dosing strategies of echinocandin drugs might provide a better efficacy in the treatment of fungal infections as compared to the current label dosing strategy. Before conducting a controlled efficacy trial of echinocandins in haematology patients, the pharmacokinetics of these alternate dosing strategies need to be tested before bringing this idea to practice in a large randomised trial.

Therefore we want to conduct a pharmacokinetic study with anidulafungin given every 48 hours or every 72 hours. This research can be performed best in a group of patients at high risk for developing invasive fungal infections.

Recipients of an allogeneic haematopoietic stem cell transplant (HSCT) or patients receiving intensive chemotherapy for acute myeloid leukaemia (AML) or myelodysplastic syndrome (MDS) are at a relatively high risk of developing invasive fungal infections and are therefore candidates for primary prophylaxis. However, the options are limited to fluconazole which affords no protection against mould infections. Amphotericin B is not considered useful because of its desoxycholate formulation has too many side effects and its lipid formulations are too expensive nor have the broad-spectrum triazoles itraconazole and voriconazole proved their value in this setting. Anidulafungin is the first of a new class of antifungal drugs quite unlike any others attacking specifically the ß 1-3 -D-glucan synthase of the cell wall. It has relatively few side effects and appears safe and effective for treating Aspergillus and Candida infections. Since these two genera account for 90% of fungal infections in HSCT recipients the drug would seem an ideal candidate for prophylaxis.

Importantly, nothing is known about the pharmacokinetics of alternate dosing regimens of anidulafungin in this patient population. Therefore a pharmacokinetic study of a homogenous cohort of patients is necessary to test the assumption, that adequate exposure is obtained with alternate dosing and that it is safe.

ELIGIBILITY:
Inclusion Criteria:

* Patient receives an allogeneic haematopoietic stem cell transplant following myeloablative chemotherapy or receives intensive chemotherapy for AML-MDS
* Subject is at least 18 and not older than 65 years of age on the day of the first dosing
* Has no signs or symptoms of invasive fungal disease
* If a woman, is neither pregnant nor able to become pregnant and is not nursing an infant
* Has an ALAT, ALAT, alkaline phosphatase < 5 times the upper limit of normal and a bilirubin level < 3 times the upper limit of normal
* Is not known to be hypersensitive to echinocandin antifungal agents
* Is managed with a quadruple central venous catheter (Arrow-Howes™ Quad-Lumen 8.5,5 French; Arrow International)
* Subject is able and willing to sign the Informed Consent before screening evaluations

Exclusion Criteria:

* Documented history of sensitivity to medicinal products or excipients similar to those found in the anidulafungin preparation
* Known of Positive HIV test or hepatitis B or C test in history
* History of QT time prolongation
* History of or current abuse of drugs, alcohol or solvents
* Inability to understand the nature of the trial and the procedures required
* Has not previously participated in this trial

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2010-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics | two weeks per subject
  comparison of pharmacokinetics of anidulafungin given once in every two days or once in every three days

SECONDARY OUTCOMES:
adequate exposure | 2 weeks for each subject; analysis after 3 months after last subject inclusion
  To determine whether adequate exposure is attained by patients undergoing an allogeneic haematopoietic stem cell transplant following myeloablative chemotherapy or receiving intensive chemotherapy for AML-MDS when using a q48 hour or a q72 hour dosing regimen
safety | 3 weeks
  To determine the safety of anidulafungin in the patient population

CONTACTS AND LOCATIONS:
Overall Officials: R Brüggemann, PharmD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Result] Bruggemann RJ, Van Der Velden WJ, Knibbe CA, Colbers A, Hol S, Burger DM, Donnelly JP, Blijlevens NM. A rationale for reduced-frequency dosing of anidulafungin for antifungal prophylaxis in immunocompromised patients. J Antimicrob Chemother. 2015 Apr;70(4):1166-74. doi: 10.1093/jac/dku477. Epub 2014 Dec 3. PMID 25473029